CLINICAL TRIAL: NCT03141463
Title: Immune Modulating Effects and Safety of Vvax001, a Therapeutic Semliki Forest Virus Based Cancer Vaccine, in Patients With a History of (Pre) Malignant Cervical Lesions.
Brief Title: Vvax001 Cancer Vaccine in (Pre) Malignant Cervical Lesions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Dutch Cancer Society (Other); ViciniVax B.V (Unknown)
Responsible Party: Principal Investigator, Refika Yigit, MD PhD, University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Vvax001-UMCG-01; 2015-004979-74 (EudraCT Number); NL56680.000.16 (Other: CCMO)
Record Dates: First submitted 2017-03-16; First posted 2017-05-05 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2017-11

CONDITIONS: CIN 2/3; Cervical Cancer
Keywords: Therapeutic vaccination
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vvax001 therapeutic cancer vaccine (Experimental): Patients will receive three consecutive doses of Vvax001, with an interval of 3 weeks
  Interventions: Biological: Vvax001 therapeutic cancer vaccine

INTERVENTIONS:
Biological: Vvax001 therapeutic cancer vaccine — Vvax001 is a vaccine consisting of a replication-incompetent Semliki Forest Virus (SFV) vector encoding HPV-derived tumor antigens. Patients will receive three consecutive doses, with an interval of 3 weeks.
  Other Names: rSFVeE6,7

SUMMARY:
Immune modulating effects and safety of Vvax001; different dosages will be tested in patients with a history of (pre) malignant cervical lesions.

DETAILED DESCRIPTION:
Vvax001 is a therapeutic cancer vaccine consisting of a replication-incompetent Semliki Forest Virus (SFV) vector encoding HPV-derived tumor antigens. Patients will receive three consecutive doses, with an interval of 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* A history of CIN II and III OR cervical cancer
* Minimally 12 weeks after completion of treatment
* Age of 18 years and older
* Baseline laboratory findings; adequate hepatic, renal ,and bone marrow function, HIV- and HBV-negative
* Patients of child-bearing potential should test negative using a serum pregnancy test and agree to utilize effective contraception during the entire treatment and follow-up period of the study
* Written informed consent according to local guidelines

Exclusion Criteria:

* Prior treatment with immunotherapeutic agents against HPV
* History of an autoimmune disease or other systemic intercurrent disease that might affect the immunocompetence of the patient, or current or prior use (4 weeks before start of the study) of high dose immunosuppressive therapy.
* History of a second malignancy except curatively treated low-stage tumors with a histology that can be differentiated from the cervical cancer type
* Participation in a study with another investigational drug within 30 days prior to the enrolment in this study
* Any condition that in the opinion of the investigator could interfere with the conduct of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-01-13 (Actual); Primary Completion 2017-11-28 (Actual); Study Completion 2017-11-28 (Actual)

PRIMARY OUTCOMES:
Immunogenicity | Day 28-31 and day 49-52 after first administration of Vvax001
  To assess the immunological activity of Vvax001 by monitoring HPV-16 E6,7-specific T-cell immune responses

SECONDARY OUTCOMES:
Number of treatment-related adverse events as assessed by CTCAE v4.0 | up to 49-52 days after first administration of Vvax001
  To monitor the side effects/ adverse events related to intramuscular administration of Vvax001. Toxicity will be graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: R Yigit, MD PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Background] Daemen T, Riezebos-Brilman A, Regts J, Dontje B, van der Zee A, Wilschut J. Superior therapeutic efficacy of alphavirus-mediated immunization against human papilloma virus type 16 antigens in a murine tumour model: effects of the route of immunization. Antivir Ther. 2004 Oct;9(5):733-42. PMID 15535411
- [Background] Riezebos-Brilman A, Walczak M, Regts J, Rots MG, Kamps G, Dontje B, Haisma HY, Wilschut J, Daemen T. A comparative study on the immunotherapeutic efficacy of recombinant Semliki Forest virus and adenovirus vector systems in a murine model for cervical cancer. Gene Ther. 2007 Dec;14(24):1695-704. doi: 10.1038/sj.gt.3303036. Epub 2007 Oct 11. PMID 17928874
- [Background] Draghiciu O, Boerma A, Hoogeboom BN, Nijman HW, Daemen T. A rationally designed combined treatment with an alphavirus-based cancer vaccine, sunitinib and low-dose tumor irradiation completely blocks tumor development. Oncoimmunology. 2015 May 27;4(10):e1029699. doi: 10.1080/2162402X.2015.1029699. eCollection 2015 Oct. PMID 26451295